CLINICAL TRIAL: NCT02229422
Title: A Study of Obinutuzumab in Combination With High-Dose Methylprednisolone in Chronic Lymphocytic Leukemia Patients
Brief Title: A Study of Obinutuzumab(GA101) in Combination With High-Dose Methylprednisolone(HDMP) in Chronic Lymphocytic Leukemia(CLL) Patients (GA101 & HDMP)
Acronym: GA101 & HDMP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas Kipps, Associate Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140396
Record Dates: First submitted 2014-08-27; First posted 2014-09-01 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: CLL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GA101/HDMP (Experimental): All subjects will receive GA101 - Obinutuzumab by IV infusion for up to 6 cycles (28-day cycles) as follow:
  * On Cycle 1, Day 1, 100 mg GA101-obinutuzumab will be administered.
  * On Cycle 1, Day 2, 900 mg of GA101-obinutuzumab will be administered.
  * On Cycle 1, Days 8 and 15, 1,000 mg of GA101-obinutuzumab will be administered.
  * On Cycles 2-6, Day 1, 1,000 mg of GA101-obinutuzumab will be administered.
  All subjects will receive HDMP by IV infusion for up to 4 cycles (28-day cycles) as follow:
  •On Cycle 1-4, Days 1 to 3, 1,000 mg/m2 Methylprednisolone will be administered.
  Interventions: Drug: GA101/HDMP

INTERVENTIONS:
Drug: GA101/HDMP — All subjects will receive GA101 - Obinutuzumab by IV infusion for up to 6 cycles (28-day cycles) as follow:
  * On Cycle 1, Day 1, 100 mg GA101-obinutuzumab will be administered.
  * On Cycle 1, Day 2, 900 mg of GA101-obinutuzumab will be administered.
  * On Cycle 1, Days 8 and 15, 1,000 mg of GA101-obinutuzumab will be administered.
  * On Cycles 2-6, Day 1, 1,000 mg of GA101-obinutuzumab will be administered.
  All subjects will receive HDMP by IV infusion for up to 4 cycles (28-day cycles) as follow:
  •On Cycle 1-4, Days 1 to 3, 1,000 mg/m2 Methylprednisolone will be administered.

SUMMARY:
We hypothesize that GA101 - Obinutuzumab in combination with HDMP is well tolerated and will induce similar if not higher response rates than the ones observed in Rituximab plus HDMP studies (Castro et al., 2009, Castro et al., 2008).

DETAILED DESCRIPTION:
This is an open label phase Ib/II clinical trial to determine the safety and clinical activity of the GA101 - Obinutuzumab in combination with high-dose methylprednisone (HDMP). We will evaluate dose-limiting toxicities (DLTs) during the first month of therapy as part of the phase Ib of this study. In the phase II we will determine response rate in an intention to treat analysis. In this study we will include CLL patients that have never received treatment as well as patients that have failed previous treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL
2. Indication for treatment as defined by the IWCLL Guidelines (Hallek et al., 2008b).
3. Males and females 18 years of age and older.
4. Laboratory parameters as specified below:

   * Hematologic: Hemoglobin > 8 g/dL (may be post-transfusion); platelet count > 40 x103/mm3 (may be post-transfusion). Absolute neutrophil count > 1.0 109 cells/mm3 (Growth factor use is allowed).
   * Hepatic: Total Bilirubin < 3 x ULN, and ALT and AST < 3 x ULN
   * Renal: Creatinine clearance > 30 mL/min (Calculated according to institutional standards or using Cockcroft-Gault formula. Subjects with requirement of hemodialysis will be excluded).
5. ECOG Performance Status < 2, unless the decline of the performance status is considered to be related to CLL symptoms.
6. Anticipated survival of at least 6 months.
7. Subjects can be enrolled and treated under this protocol regardless of their CLL treatment history or number of previous treatments. In addition, subjects with history of allogeneic stem cell transplant can be enrolled and treated unless they have active manifestations of graft vs. host disease (GVHD) or chronic illness or infections that will prevent them from completing the study.
8. Previously untreated subjects that meet ANY of the following criteria: A. Documented refusal to be treated with chemotherapy agents. B. Subjects that are not candidates for treatment with chemotherapy based on poor performance status (ECOG ≥ 2), advance age (> 65 years), Cumulative Illness Rating Scale (CIRS score) ≥ 6 or cytopenias.
9. Effective contraception is required while receiving GA101 - Obinutuzumab. For women of childbearing potential and men, effective contraception is required while receiving GA101 - Obinutuzumab and for 365 days (12 months) after the last dose of the study drug.
10. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
11. Subjects must give written informed consent to participate in this trial.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Treatment with chemotherapy, monoclonal antibodies or biological agents (e.g. Ibrutinib, lenalidomide) within 28 days prior to entering the study.
3. Treatment with chemotherapy, monoclonal antibodies, biological agents (e.g. Ibrutinib) or other than the investigational agents during the time of participation in this trial.
4. Grade 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
5. Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, COPD)
6. Participation in any investigational drug study within 28 days prior to initiation of treatment within this protocol.
7. History of second malignancy, other than non-melanoma skin cancer or in situ carcinoma of the cervix or the breast, unless the tumor was successfully treated at least 2 years before trial entry and with no evidence of relapse or active cancer.
8. Active symptomatic fungal, bacterial and/or viral infection including evidence of infection with HIV, human T-cell leukemia virus 1 (HTLV-1) seropositive status.
9. Evidence of active acute or chronic Hepatitis B (HBV).
10. Evidence of active Hepatitis C (HCV): subjects with positive hepatitis C serology AND positive HCV RNA test.
11. Any illness or condition that in the opinion of the Investigator may affect safety of treatment or evaluation of any the study's endpoints.
12. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
13. Known hypersensitivity to any of the study drugs.
14. Major surgery (within 4 weeks prior to the start of Cycle 1), except for procedures that are performed for diagnostic purposes.
15. Men or women of childbearing potential who refuse to use an adequate measure of contraception (oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly) unless they have past medical history of surgical sterilization.
16. Vaccination with a live vaccine within 28 days of the initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Adverse events that constitute the Dose Limiting Toxicity | 2 months
Response assessment based on IWCLL | 2 months

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
Overall Survival and Minimal residual disease (MRD) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kipps Thomas, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States